CLINICAL TRIAL: NCT05814302
Title: Treatment Of Fever And Associated Symptoms In The Emergency Department: Which Drug To Choose?
Brief Title: Treatment Of Fever In The Emergency Department
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3710
Record Dates: First submitted 2023-02-14; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-02

CONDITIONS: Fever
Keywords: Fever; Paracetamol; Paracetamol/Ibuprofen; Emergency Department
MeSH Terms: conditions — Fever; Emergencies | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Paracetamol — Emergency physicians were free to administer paracetamol 1000 mg (P), the combination paracetamol 500 mg/ibuprofen 150 mg (PI) or Ibuprofen 600 mg (I)
  Other Names: Combination of paracetamol/ibuprofen

SUMMARY:
Fever is a frequent cause of admission to the Emergency Department (ED) around the world. While it can be caused by a wide range of conditions, the most effective treatment based on its etiology is still undetermined. This observational, prospective, single-center study enrolled adult patients who accessed the ED for fever, with the aim to define the most effective treatment for them.

DETAILED DESCRIPTION:
Physicians were free to administer paracetamol 1000 mg (P), the combination paracetamol 500 mg/ibuprofen 150 mg (PI) or Ibuprofen 600 mg (I).The primary endpoint was both 1-degree and 1-point reduction in body temperature for all associated symptoms on the Numeric Rating Scale (NRS) after 1 hour (T1). Secondary endpoint was the reduction of at least 2 points on the NRS after two hours (T2). Adverse events, the needing of a rescue therapy and the response based on the underlying etiology (bacterial, viral, or immune/neoplastic) were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* fever with/without associated symptoms
* adults who had given their consent to participate in the study.

Exclusion Criteria:

* age < 18 years old
* contraindications or allergies to Paracetamol, Ibuprofen or to the combination Paracetamol/Ibuprofen
* patients unable to take oral drugs
* patients who did not express their consent to participate to the study

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults > 18 years old with fever and associated symptoms accessing the ED
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
body temperature | 1 hour
  the reduction of 1-degree of body temperature after 1 hour (T1) after the drug administration
Numerical Rating Scale (NRS) | 1 hour
  the reduction of 1-point for all associated symptoms on NRS after 1 hour (T1) after the drug administration. NRS is a "0-10" scale tool to assess pain severity, with zero that means "no pain" and 10 "the worst pain".

SECONDARY OUTCOMES:
the reduction of at least 2 points on the Numerical Rating Scale (NRS) after two hours (T2) after the drug administration | 2 hours
  the secondary endpoint was to evaluate the number of patients (%) who obtained a reduction of at least 2 points on the NRS scale, in at least one of the symptoms associated with fever 2 hours after the antypiretic administration (T2). NRS is a "0-10" scale tool to assess pain severity, with zero that means "no pain" and 10 "the worst pain".
rescue therapy | 2 hours
  to identify the number of patients (%) who needed a rescue therapy
adverse events | 2 hours
  to identify the percentage (%) of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Roma, Italy